CLINICAL TRIAL: NCT01338753
Title: A Multicenter Phase II Study, to Evaluate the Predictive Markers of Response in Locally Advanced Breast Cancer, Treated With Bevacizumab Combined With Neoadjuvant Chemotherapy
Brief Title: Study to Evaluate Markers of Response in Locally Advanced Breast Cancer
Acronym: IMAGING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ML22197/2009-01; 2009-011037-27 (EudraCT Number)
Record Dates: First submitted 2011-03-04; First posted 2011-04-19 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Breast Neoplasms
Keywords: breast; cancer; Pharmacogenomics; bevacizumab
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Bevacizumab; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Bevacizumab, docetaxel and doxorubicin followed by surgery — The dosage form is Parenteral Injection (I/V) for all study drugs. Bevacizumab 15mg/kg in a single dose on day 1. Then 3 weeks later begin the cycles. On the day 1 of the cycle the patient receives Bevacizumab 15mg/kg, docetaxel 60mg/m2 and doxorubicin 50mg/m2.
  The cycles have a frequency of one every three weeks, and the protocol defines 4 cycles in total.
  The surgical procedure will be done 4-6 weeks after completion of chemotherapy.
  Other Names: Avastin; Taxotere; Adriamycin

SUMMARY:
The purpose of this study is to compare the association between image and certain molecular markers with complete response in patients with locally advanced breast cancer, treated with neoadjuvant chemotherapy composed of Bevacizumab, Docetaxel and Doxorubicin.

DETAILED DESCRIPTION:
This is a pharmacogenomic phase II, multicenter, prospective clinical trial whose main objective is to evaluate the association of molecular and imaging markers with the response to bevacizumab administration in combination with docetaxel and doxorubicin as neoadjuvant chemotherapy in patients diagnose with locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Signed Informed consent form
* Ages between 18 and 70
* 12 months of life expectancy at least
* Histologically confirmed breast cancer
* No previous treatment for locally advanced breast cancer
* Her2+ o Her2-
* Disease measurable by PET and/or MRI
* ECOG 0-1
* Adequate organic function
* Negative pregnancy test; fertile women must use anticonceptive methods after ICF and 30 days after last study drug administration
* Enough capability to follow the procedures and follow-up test included in the protocol

Exclusion Criteria:

* Metastatic disease
* Inadequate health to receive the study chemotherapy
* Previous breast cancer treatment
* Pregnant or lactating women
* Major surgery or significative traumatic injure in the 28 days previous to inclusion, or during treatment.
* Minor surgery 24 hours before first bevacizumab infusion
* Concomitant or recent aspirin(>325mg/day)or clopidogrel(>75mg/day) treatment
* Concomitant or recent oral anticoagulant treatment
* History or evidence or bleeding diathesis or hereditary coagulopathy with bleeding risk
* Uncontrolled arterial hypertension
* Clinical significative heart disease, or uncontrolled severe arrhythmia disorder
* Unhealed wounds, peptic ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intrabdominal abscess, 6 months before inclusion
* Evidence of any other disease, neurological or metabolical disorder or physical examination or laboratory finding related with any disease that makes the subjet ineligible for the study treatment or that put the subject in risk because of the study treatment.
* Psychiatric disorders that may prevent the subject to complete the study treatment
* Current participation in any other trial involving an investigational drug, or participation in any kind of trial 28 days before inclusion
* Chronical corticosteroid treatment
* Hypersensitivity reaction to bevacizumab or any of its components or any of the other study drugs or components
* Patients diagnosed with different neoplasms the previous 5 years excluding non melanoma skin cancer and resected cervical cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of SNPs genotyping. | This evaluation will be performed within 14 days before start of treatment
  The analysis of genetic differences will be determined through analysis of single nucleotide polymorphisms. It will be assesed before starting the treatment using Affymetrix's Human Mapping 500k array set.
Assessment of tumoral response by Dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) | This evaluation will be performed within 14 days before start of treatment (baseline assesment).
  The radiological interpretation of the images will evaluate size, shape, extent, distribution and kinetics of the lesons according to American College of Radiology Breast Imaging Reporting and Data System (ACR BIRADS- MRI (2003) guidelines).
Assessment of tumoral response by Dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) | This evaluation will be performed within 12-19 days after first cycle
  The radiological interpretation of the images will evaluate size, shape, extent, distribution and kinetics of the lesons according to American College of Radiology Breast Imaging Reporting and Data System (ACR BIRADS- MRI (2003) guidelines).
Assessment of tumoral response by Dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) | This evaluation will be performed within 12-19 days aftet fifth cycle.
  The radiological interpretation of the images will evaluate size, shape, extent, distribution and kinetics of the lesons according to American College of Radiology Breast Imaging Reporting and Data System (ACR BIRADS- MRI (2003) guidelines).
Positron emission tomography (PET) scan | This evaluation will be performed within 14 days before start of treatment (baseline assesment)
  It will be determined the association between tissue:blood activity ratio and hypoxic tumor volume by 18F-fluoromisonidazole positron emission tomography (FMISO-PET). DNA synthesis, assesed by [18F]-fluoro-3'-deoxy-3'-L-fluorothymidine PET (FLT-PET), will be compared to quantitative kinetics data adquired through previously described DCE-MRI. Finally, these results will be correlated with the Risk Score obtained in the genomic analysis
Positron emission tomography (PET) scan | This evaluation will be performed within 12-19 days after first cycle
  It will be determined the association between tissue:blood activity ratio and hypoxic tumor volume by 18F-fluoromisonidazole positron emission tomography (FMISO-PET). DNA synthesis, assesed by [18F]-fluoro-3'-deoxy-3'-L-fluorothymidine PET (FLT-PET), will be compared to quantitative kinetics data adquired through previously described DCE-MRI. Finally, these results will be correlated with the Risk Score obtained in the genomic analysis
Positron emission tomography (PET) scan | This evaluation will be performed within 12-19 days aftet fifth cycle
  It will be determined the association between tissue:blood activity ratio and hypoxic tumor volume by 18F-fluoromisonidazole positron emission tomography (FMISO-PET). DNA synthesis, assesed by [18F]-fluoro-3'-deoxy-3'-L-fluorothymidine PET (FLT-PET), will be compared to quantitative kinetics data adquired through previously described DCE-MRI. Finally, these results will be correlated with the Risk Score obtained in the genomic analysis
Evaluation of Genomic tissular profile in a sample of biopsy | This evaluation will be performed within 14 days before start of treatment (baseline assesment
  A correlative analysis will be performed between the expression profile of the sample obtained by Affymetrix 's GeneChip Human Genome U133 and its association with tumor response (based on the imaging markers described previously) on the proposed stages (baseline, before first cycle of treatment and after fifth cycle of treatment
Evaluation of Genomic tissular profile in a sample of biopsy | This evaluation will be performed within 12-19 days after first cycle
  A correlative analysis will be performed between the expression profile of the sample obtained by Affymetrix 's GeneChip Human Genome U133 and its association with tumor response (based on the imaging markers described previously) on the proposed stages (baseline, before first cycle of treatment and after fifth cycle of treatment
Evaluation of Genomic tissular profile in a sample of biopsy | This evaluation will be performed within 12-19 days aftet fifth cycle
  A correlative analysis will be performed between the expression profile of the sample obtained by Affymetrix 's GeneChip Human Genome U133 and its association with tumor response (based on the imaging markers described previously) on the proposed stages (baseline, before first cycle of treatment and after fifth cycle of treatment).
Evaluation of Proteomic expression in blood serum | This evaluation will be performed within 14 days before start of treatment (baseline assesment)
  To determine the proteomic expression in blood serum, a ZeptoMARK Reverse Array assay will be performed according to manufacturer's instructions.
Evaluation of Proteomic expression in blood serum | This evaluation will be performed within 12-19 days after first cycle. Description:
  To determine the proteomic expression in blood serum, a ZeptoMARK Reverse Array assay will be performed according to manufacturer's instructions.
Evaluation of Proteomic expression in blood serum | This evaluation will be performed within 12-19 days aftet fifth cycle.
  To determine the proteomic expression in blood serum, a ZeptoMARK Reverse Array assay will be performed according to manufacturer's instructions.

SECONDARY OUTCOMES:
Evaluation of Complete pathological response in surgical piece | This evaluation will be performed within 20-22 weeks after start of treatment.
  To determine if a patient has undergone complete pathological response, an anatomo-pathological study will be conducted on the surgical piece. The evaluation will follow the Miller and Payne criteria; a complete response will be considered just in the absence of invasive tumor cells in breast and lymphatic nodules.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Anton, MD, Principal Investigator — Hospital Miguel Servet; Jesus Garcia-Foncillas, MD, Principal Investigator — Clinica Universitaria de Navarra; Alfonso Yubero, MD, Principal Investigator — Hospital Obispo Polanco; Isabel Alvarez, MD, Principal Investigator — Hospital Donosti; Jose Manuel Lopez-Vega, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Blanca Hernando, MD, Principal Investigator — Hospital General Yagüe; Jose Juan Illarramendi, Md, Principal Investigator — Hospital de Navarra; Irene Gil, MD, Principal Investigator — Hospital de Tudela; Purificacion Martinez del Prado, MD, Principal Investigator — Hospital de Basurto; Rosa Sanchez, MD, Principal Investigator — Complejo Hospitalario San Millán San Pedro De La Rioja; Arrate Plazaola, MD, Principal Investigator — Onkologikoa; Serafin Morales, MD, Principal Investigator — Hospital Universitario Arnau Vilanova de Lleida
Locations (11):
- Spain (11):
  - Hospital Obispo Polanco, Teruel, Aragon
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital General Yagüe, Burgos, Burgos
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital de Donosti, San Sebastián, Guipúzcoa
  - Onkologikoa, San Sebastián, Guipúzcoa
  - Hospital de San Millan, Logroño, La Rioja
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital de Tudela, Tudela, Navarre
  - Hospital de Basurto, Bilbao, Vizcaya